CLINICAL TRIAL: NCT03859986
Title: A Phase 2, Randomized, Double-Blind, Vehicle-Controlled, Parallel-Group Study To Evaluate The Safety And Efficacy Of ALX-101 Topical Gel Administered Twice Daily In Adult And Adolescent Subjects With Moderate Atopic Dermatitis
Brief Title: Study in Subjects With Moderate Atopic Dermatitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ralexar Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALX-101-ATOP-204
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Atopic Dermatitis Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALX-101 Gel 5% (Experimental): ALX-101 Gel 5% applied topically twice daily for 56 days
  Interventions: Drug: ALX-101 Gel 5%
- ALX-101 Gel Vehicle (Placebo Comparator): ALX-101 Gel Vehicle applied topically twice daily for 56 days
  Interventions: Drug: ALX-101 Gel Vehicle

INTERVENTIONS:
Drug: ALX-101 Gel Vehicle — ALX-101 Gel Vehicle
  Arms: ALX-101 Gel Vehicle
Drug: ALX-101 Gel 5% — ALX-101 Gel 5%
  Arms: ALX-101 Gel 5%

SUMMARY:
This is a Phase 2, randomized, double-blind, vehicle-controlled, parallel-group study to evaluate the safety and efficacy of ALX-101 Gel 5% and a matching ALX-101 Gel Vehicle when applied topically twice daily for 56 days in adult and adolescent subjects with moderate atopic dermatitis

DETAILED DESCRIPTION:
The main objectives of this study are to:

* Evaluate the safety of ALX-101 Gel 5% when applied topically twice daily in subjects with moderate atopic dermatitis compared with a matching ALX-101 Gel Vehicle
* Evaluate the efficacy of ALX-101 Gel 5% when applied topically twice daily in subjects with moderate atopic dermatitis compared with a matching ALX-101 Gel Vehicle

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 12 years of age at the time of consent.
2. Subject has a clinical diagnosis of stable AD confirmed using the Hanafin and Rajka criteria
3. Subject has at least a 6-month history of atopic dermatitis and had no significant flares in atopic dermatitis for at least 4 weeks before Visit 1 (screening) (information obtained from medical chart or subject's physician or directly from the subject).
4. Subject must have active features of AD covering a minimum of 2% body surface area (BSA) (excluding scalp, face, genitals, palmar aspect of hands and plantar aspect of feet) at Visit 2 (baseline).
5. Subject has moderate AD, defined as vIGA-AD™ score of 3 ("moderate"), at Visit 2 (baseline).
6. Subject has an EASI score ≥ 5 at Visit 2 (baseline)
7. Subject has been using an emollient (except those containing urea) daily for at least 1 week prior to Visit 2 (baseline), except on visit day before the visit. Subject agrees to continue using that emollient, daily at the same frequency, on non-treated areas, throughout the study but not the day of visits prior to the visit scheduled time.
8. Female subject of childbearing potential involved in any sexual intercourse that could lead to her pregnancy, must have a negative serum pregnancy test at Visit 1, a negative urine pregnancy test at Visit 2 (baseline) and agree to use an approved highly effective contraceptive method for the entire study and up to 4 weeks following the final dose of study medication unless they are surgically sterile (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy) or in menopausal state for at least one year prior to screening (Visit 1)
9. Male subject of childbearing potential agree to use an approved highly effective method of contraception through study participation for 4 weeks following the final dose of study medication
10. Subject is in good general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair evaluation of the AD being treated or which exposes the subject to an unacceptable risk by study participation
11. Subject is willing and able to follow all study instructions and to attend all study visits
12. Subject is able to comprehend and willing to sign an Informed Consent Form (ICF)/Assent Form (AF)
13. Parent/guardian has the ability to understand, agree to and sign the study Informed Consent Form (ICF) prior to initiation of any protocol-related procedures as applicable; subject has the ability to give assent in the Assent Form (AF)
14. Informed Consent Form (ICF)/Assent Form (AF) must be obtained prior to initiation of any protocol-related procedures.

Exclusion Criteria:

1. Subject has spontaneously improving or rapidly deteriorating AD
2. Subject has clinically infected AD
3. Subject has any signs or symptoms associated with topical AD therapy which, in the investigator's opinion, might impair evaluation of the AD being treated or which exposes the subject to an unacceptable risk by study participation
4. Subject has any clinically significant laboratory abnormality, medical condition or physical/vital signs abnormality that would, in the opinion of the investigator, put the subject at undue risk or interfere with interpretation of study results
5. Subjects with a past history of cancer or lymphoproliferative disease within 5 years prior to Visit 2 (baseline) (subjects with successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix are not to be excluded)
6. Subject is known to have immune deficiency or is immunocompromised
7. Subject has a known history of chronic infectious disease (e.g., hepatitis B, hepatitis C, or infection with human immunodeficiency virus)
8. Subject had major surgery within 8 weeks prior to Visit 2 (baseline) or has a major surgery planned during the study.
9. Topical medications, including but not limited to, topical corticosteroids, crisaborole and any other topical phosphodiesterase-4 inhibitor, calcineurin inhibitors, tars, bleach, antimicrobials, medical devices and bleach bath within 2 weeks prior to Visit 2 (baseline)
10. Subject has used any non-medicated topical product (e.g., lotions, gels, creams, ointments) in the planned treatment area 4 hours prior to Visit 2 (baseline)
11. Subject has used the following systemic treatments (other than biologics) that could affect atopic dermatitis less than 4 weeks prior to Visit 2 (baseline) (e.g., retinoids, calcineurin inhibitors, methotrexate, cyclosporine, hydroxycarbamide [hydroxyurea], azathioprine, oral/injectable corticosteroids) within 4 weeks prior to Screening. Intranasal corticosteroids and inhaled corticosteroids are allowed. Eye and ear drops containing corticosteroids are also allowed.
12. Subject has used any systemic antibiotics within 2 weeks prior to Visit 2 (baseline)
13. Subject has used hydroxyzine or diphenhydramine within 1 week prior to Visit 2 (baseline), unless on a stable dose.
14. Subject has used topical doxepin within 1 week prior to Visit 2 (baseline).
15. Subject has used topical products containing urea within 1 week prior to Visit 2 (baseline)
16. Subject has used or is planning to use any phototherapy (e.g., UVA/UVB therapy, or PUVA therapy), excessive natural or artificial ultraviolent radiation (e.g., sunlight, tanning beds) which, in the investigator's opinion, might affect AD within 4 weeks prior to Visit 2 (baseline)
17. Biologic therapies (e.g., Dupilumab) within 12 weeks or 5 half-lives prior to Visit 2 (baseline)
18. Subject has a history of sensitivity to any of the ingredients in the study medications
19. Subject has any known concomitant dermatologic or medical condition which, in the investigator's opinion, might impair evaluation of the areas of AD being treated or which exposes the subject to an unacceptable risk by study participation (e.g., psoriasis, rosacea, lichen planus, lichen simplex chronicus,…)
20. Subject is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the study.
21. Subject has a known history of clinically significant drug or alcohol abuse in the last year prior to Visit 2 (baseline)
22. Subject has participated in a nonbiological investigational drug trial in which administration of an investigational study medication occurred within 4 weeks prior to Visit 2 (baseline)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Eczema Area Severity Index (EASI) | Day 57
  Mean change from baseline in EASI score at Week 8

CONTACTS AND LOCATIONS:
Locations (22):
- United States (20):
  - Ralexar Investigational Site 10, Beverly Hills, California
  - Ralexar Investigational Site 5, Los Angeles, California
  - Ralexar Investigational Site 3, Aventura, Florida
  - Ralexar Investigational Site 2, Jacksonville, Florida
  - Ralexar Investigational Site 22, Miami, Florida
  - Ralexar Investigational Site 18, Pinellas Park, Florida
  - Ralexar Investigational Site 6, Sanford, Florida
  - Ralexar Investigational Site 13, Marietta, Georgia
  - Ralexar Investigational Site 7, Boise, Idaho
  - Ralexar Investigational Site 21, Gurnee, Illinois
  - Ralexar Investigational Site 1, Indianapolis, Indiana
  - Ralexar Investigational Site 17, Louisville, Kentucky
  - Ralexar Investigational Site 12, Las Vegas, Nevada
  - Ralexar Investigational Site 14, Beachwood, Ohio
  - Ralexar Investigational Site 8, Fairborn, Ohio
  - Ralexar Investigational Site 9, Oklahoma City, Oklahoma
  - Ralexar Investigational Site 19, Spartanburg, South Carolina
  - Ralexar Investigational Site 16, Austin, Texas
  - Ralexar Investigational Site 4, San Antonio, Texas
  - Ralexar Investigational Site 15, Seattle, Washington
- Canada (2):
  - Ralexar Investigational Site 20, Toronto, Ontario
  - Ralexar Investigational Site 11, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided